CLINICAL TRIAL: NCT07109648
Title: Evaluating the Impacts of a Well-Being Mobile App in Mexico
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00006401; SA24-03-08 (Other Grant/Funding Number: GDI Solutions, Inc)
Record Dates: First submitted 2025-07-24; First posted 2025-08-07 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-07

CONDITIONS: Mental Health; Wellbeing
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Participants do not have access to the app during the study.
- Access to app (Experimental): Participants will be offered free premium access to the app for three months
  Interventions: Behavioral: Access to app

INTERVENTIONS:
Behavioral: Access to app — The intervention is offering a free subscription to a mental health app that combines self-guided digital tools with AI-powered support. The app features functions such as an emotional diary and structured courses on topics including managing anxiety and stress regulation. A personalized chatbot, powered by large language models (LLMs) and trained on content grounded in cognitive behavioral therapy, delivers evidence-based strategies such as cognitive restructuring, behavioral activation, and emotion regulation. The chatbot also guides users through these resources using natural, supportive conversations.
  Participants were randomly assigned to one of two groups:
  A treatment group offered free access to the app for three months, or A control group, which will receive free access to the app for one month at the end of the study
  Arms: Access to app

SUMMARY:
The researchers will study the impacts of offering access to an emotional well-being phone app to women in psychological distress in Mexico. The primary outcome is participants' psychological well-being and mental health.

ELIGIBILITY:
Inclusion Criteria:

* PHQ-4 scale equal or greater than 3
* Access to a smartphone and whatsapp
* Less than graduate school education
* Leaves in Mexico
* Earn less than 26,000 Mexican pesos

Exclusion Criteria:

* If she doesn't meet any of the inclusion criteria

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 4000 (Estimated)
Dates: Start 2023-04-18 (Actual); Primary Completion 2025-08-15 (Estimated); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
Wellbeing | From enrollment to 3 and 8 weeks after
  Measured using the World Health Organization-Five Well-Being Index (who-5). The raw score ranges from zero to 25, zero representing worst possible mental well-being and 25 representing best possible mental well-being.
Anxiety | From enrollment to 3 and 8 weeks after
  Measured using General Anxiety Disorder-7 scale (GAD-7). This is calculated by assigning scores of 0, 1, 2, and 3 to the response categories, respectively, of "not at all," "several days," "more than half the days," and "nearly every day." GAD-7 total score for the seven items ranges from 0 to 21. The definitions are:
  0-4: minimal anxiety (better outcome) 5-9: mild anxiety 10-14: moderate anxiety 15-21: severe anxiety (worse outcome)
Depression | From enrollment to 3 and 8 weeks after
  Mesured using Personal Health Questionnaire Depression Scale (PHQ-8). This is calculated by assigning scores of 0, 1, 2, and 3 to the response categories, respectively, of "not at all," "several days," "more than half the days," and "nearly every day." PHQ-8 total score for the eight items ranges from 0 to 24. The definitions are:
  Less than 5: Minimal depression (better outcome) 5-9: Mild depression 10-14: Moderate depression 15-19: Moderately severe depression More or equal to 20: Severe depression (worse outcome)
Stress | From enrollment to 3 and 8 weeks after
  Measured using Perceived Stress Scale 4 (PSS-4). The scores range from 0 to 16 where higher scores are correlated to more stress (worse outcome)

SECONDARY OUTCOMES:
Social media use - TikTok | At 3 and 8 weeks after enrollment
  Number of days in the last seven days the participant used TikTok

OTHER OUTCOMES:
Ongoing affect | Weekly from rectuiment up to 12 weeks.
  Measured through a purposely designed "emoji" survey, where the participants is asked how the participant is feeling. The options are very well, neutral, very bad. After it is constructed as a dummy variable that takes value of one if the participant answered "very well" or zero otherwise
Sleep quantity | At 3 and 8 weeks after enrollment
  hours slept the night before
Sleep quality | At 3 and 8 weeks after enrollment
  The number of times participants experienced sleep interruptions the night before
Social media use - Facebook | At 3 and 8 weeks after enrollment
  number of days in the last seven days the participant has used Facebook
Psychotherapy | At 3 and 8 weeks after enrollment
  If the participant visit recently a therapist
Effort | At 3 and 8 weeks after enrollment
  Performance on an incentive-compatible, real-effort task, where the participant needs to count the number of zeros in matrices of five columns and five rows where there are zeros and ones. The measure is the correct answers within one minute
Emotional interference | At 3 and 8 weeks after enrollment
  reaction time in the emotional Stroop task, specifically for matching colors of emotionally salient words.
  The emotional Stroop task is a variation of the Stroop effect that explores how emotional stimuli impact cognitive processing. Participants are presented with words in different colors and asked to name the ink color while ignoring the word's meaning. Longer reaction times for emotional words (e.g., "fear," "sadness") compared to neutral words (e.g., "table," "chair") indicate interference from the emotional content
Healthful habits | At 3 and 8 weeks of enrollment
  The index is calculated following Anderson (2008) and includes six standardized outcomes: the number of days in the last seven days the person exercised, went outside, did not miss work, did not raise her voice in anger, helped with homework, and had 10 minutes of self-time.
Isolation | At 3 and 8 weeks of enrollment
  Emotional and social isolation, measured by the Gierveld Loneliness Scale. It has a range of scores from 0 (least lonely, better outcome) to 6 (most lonely, worse outcome)
Perceptions of efficacy | At 3 and 8 weeks after enrollment
  measured using the Generalized Self-Efficacy Scale (GSE). The total score ranges between 10 and 40, with a higher score indicating more self-efficacy (better outcome).
Social media use - X | At 3 and 8 weeks after enrollment
  number of days in the last seven days the participant has used X
Social media use - Instagram | At 3 and 8 weeks after enrollment
  Number of days in the last seven days the participant used Instagram

CONTACTS AND LOCATIONS:
Locations (1):
- The University if Texas at Austin, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No